CLINICAL TRIAL: NCT02360215
Title: A Randomized Phase III Trial of Memantine and Whole-Brain Radiotherapy With or Without Hippocampal Avoidance in Patients With Brain Metastases
Brief Title: Memantine Hydrochloride and Whole-Brain Radiotherapy With or Without Hippocampal Avoidance in Reducing Neurocognitive Decline in Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRG-CC001; NCI-2015-00030 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC001 (Other: NRG Oncology); NRG-CC001 (Other: DCP); NRG-CC001 (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2020-02

CONDITIONS: Cognitive Impairment; Metastatic Malignant Neoplasm in the Brain; Solid Neoplasm
MeSH Terms: conditions — Cognitive Dysfunction; Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WBRT + Memantine (Experimental): Whole brain radiation therapy (WBRT) and memantine
  Interventions: Drug: Memantine; Radiation: Whole brain radiation therapy
- HA-WBRT/IMRT+ Memantine (Experimental): Whole brain radiation therapy with hippocampal avoidance (HA-WBRT) using intensity modulated radiation therapy (IMRT) and memantine
  Interventions: Radiation: Whole brain radiation therapy with hippocampal avoidance; Drug: Memantine

INTERVENTIONS:
Radiation: Whole brain radiation therapy with hippocampal avoidance — Intensity modulated radiation therapy (IMRT) 30 Gy in 10 fractions once per day, 5 days per week for approximately two week; starting within 21 calendar days after randomization.
  Other Names: IMRT; Intensity Modulated RT; INTENSITY-MODULATED RADIATION THERAPY; Intensity-Modulated Radiotherapy; Whole-brain radiation therapy; WBRT; whole-brain radiotherapy; HA-WBRT
  Arms: HA-WBRT/IMRT+ Memantine
Drug: Memantine — Given PO daily during and after radiation therapy for a total of 24 weeks. Week 1: 5 mg in the AM, none in the PM; Week 2: 5 mg in the AM, 5 mg in the PM; Week 3: 10 mg in the AM, 5 mg in the PM; Weeks 4-24: 10 mg in the AM, 10 mg in the PM. Should start the same day as radiation therapy, at latest before the fourth radiation treatment.
  Other Names: Ebixia; Memantine Hydrochloride; Namenda
Radiation: Whole brain radiation therapy — Whole brain radiation therapy (WBRT) 30 Gy in 10 fractions once per day, 5 days per week for approximately 2 weeks
  Other Names: WBRT; whole-brain radiation therapy; whole-brain radiotherapy
  Arms: WBRT + Memantine

SUMMARY:
This randomized phase III trial compares memantine hydrochloride and whole-brain radiotherapy with or without hippocampal avoidance in reducing neurocognitive decline in patients with cancer that has spread from the primary site (place where it started) to the brain. Whole brain radiotherapy (WBRT) is the most common treatment for brain metastasis. Unfortunately, the majority of patients with brain metastases experience cognitive (such as learning and memory) deterioration after WBRT. Memantine hydrochloride may enhance cognitive function by binding to and inhibiting channels of receptors located in the central nervous system. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Using radiation techniques, such as intensity modulated radiotherapy to avoid the hippocampal region during WBRT, may reduce the radiation dose to the hippocampus and help limit the radiation-induced cognitive decline. It is not yet known whether giving memantine hydrochloride and WBRT with or without hippocampal avoidance works better in reducing neurocognitive decline in patients with brain metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the addition of whole-brain radiotherapy with hippocampal avoidance (HA-WBRT) increases time to neurocognitive failure at months 2, 4, 6, and 12 as measured by neurocognitive decline on a battery of tests: the Hopkins Verbal Learning Test-Revised (HVLT-R) for Total Recall, Delayed Recall, and Delayed Recognition, Controlled Oral Word Association (COWA), and the Trail Making Test (TMT) Parts A and B.

SECONDARY OBJECTIVES:

I. Determine whether the addition of HA-WBRT preserves neurocognitive function at months 2, 4, 6, and 12 as separately measured by each test, the HVLT-R for Total Recall, Delayed Recall, and Delayed Recognition; COWA; and TMT Parts A and B.

II. Evaluate the potential benefit of HA-WBRT in symptom burden, as measured by the M. D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT).

III. Assessment of quality adjusted survival and cost analysis using the five-level version of the EuroQol five-dimensional (EQ-5D-5L).

IV. Compare cumulative incidence of progression and overall survival after WBRT versus HA-WBRT.

V. Compare adverse events between the treatment arms according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 criteria.

TERTIARY OBJECTIVES:

I. Collect serum, plasma, and imaging studies for future translational research analyses.

II. Evaluate magnetic resonance (MR) imaging biomarkers of white matter injury and hippocampal volumetry at baseline and 6 months as potential predictors of neurocognitive decline and differential benefit from HA-WBRT as compared to WBRT.

III. Association of symptom burden and anxiety/depression with neurocognitive function.

IV. Evaluate the potential correlation between the prognostic scoring systems Radiation Therapy Oncology Group (RTOG) recursive partitioning analysis (RPA) and the diagnosis-specific graded prognostic assessment (DS-GPA) and neurocognitive function at baseline and overtime.

After completion of study treatment, patients are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:

  * Brain metastases outside a 5-mm margin around either hippocampus must be visible on contrast-enhanced magnetic resonance imaging (MRI) performed =< 21 days prior to Step 1 registration; an allowed exception, regarding ability to image brain metastases, would be that patients who had undergone radiosurgery or surgical resection and are planning adjuvant WBRT do not have to have visible disease but do need a pre-surgery MRI or computed tomography (CT) scan demonstrating brain metastases; however, the brain metastases could not have been within 5 mm of either hippocampus
  * Patients must have a gadolinium contrast-enhanced three-dimensional spoiled gradient (SPGR), magnetization-prepared rapid gradient echo (MP-RAGE), or turbo field echo (TFE) axial MRI scan with standard axial and coronal gadolinium contrast-enhanced T1-weighted sequence and axial T2/FLAIR sequence acquisitions; to yield acceptable image quality, the gadolinium contrast-enhanced three-dimensional SPGR, MP-RAGE, or TFE axial MRI scan should use the smallest possible axial slice thickness not exceeding 1.5 mm; the associated coronal and sagittal contrast-enhanced T1 sequences can be up to 2.5 mm in slice thickness; this MRI must be obtained =< 21 days prior to step 1 registration; the vendor specific MRI protocols are available for download from the Alzheimer's Disease Neuroimaging Initiative (ADNI)
  * Patients must provide study-specific informed consent prior to registration
* PRIOR TO STEP 2 REGISTRATION:

  * The following baseline neurocognitive assessments must be completed prior to Step 2 registration: HVLT-R, TMT, and COWA;
  * Pathologically (histologically or cytologically) proven diagnosis of solid tumor malignancy within 5 years prior to Step 2 registration
  * History and physical examination within 28 days prior to Step 2 registration
  * Karnofsky performance status of >= 70 within 28 days prior to Step 2 registration
  * Serum creatinine =< 3 mg/dL (265 umol/L) and creatinine clearance >= 30 ml/min
  * Blood urea nitrogen (BUN) within institutional upper limit of normal (e.g. < 20 mg/dL)
  * Total bilirubin =< 2.5 mg/dL (43 umol/L)
  * Patients may have had prior therapy for brain metastasis, including radiosurgery and surgical resection; patients must have completed prior therapy by at least 14 days prior to Step 2 for surgical resection and 7 days for radiosurgery
  * Negative serum pregnancy test (in women of childbearing potential) =< 14 days prior to Step 2; women of childbearing potential and men who are sexually active must practice adequate contraception while on study
  * Patients who are primary English or French speakers are eligible

Exclusion Criteria:

* Prior external beam radiation therapy to the brain or whole brain radiation therapy
* Planned cytotoxic chemotherapy during the WBRT only; patients may have had prior chemotherapy
* Radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, including placement of external ventricular drain or ventriculoperitoneal shunt
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other acute respiratory illness precluding study therapy at the time of registration
  * Severe hepatic disease defined as a diagnosis of Child-Pugh class B or C hepatic disease
  * Renal tubular acidosis or metabolic acidosis
  * Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; Note also that HIV testing is not required for eligibility for this protocol
* Pregnant or lactating women, or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior allergic reaction to memantine (memantine hydrochloride)
* Current alcohol or drug abuse (may exacerbate lethargy/dizziness with memantine)
* Intractable seizures while on adequate anticonvulsant therapy-more than 1 seizure per month for the past 2 months
* Patients with definitive leptomeningeal metastases
* Patients with brain metastases from primary germ cell tumors, small cell carcinoma, unknown primary, or lymphoma
* Contraindication to magnetic resonance (MR) imaging such as implanted metal devices or foreign bodies
* Contraindication to gadolinium contrast administration during MR imaging, such as allergy or insufficient renal function
* Current use of (other N-methyl D-aspartate [NMDA] antagonists) amantadine, ketamine, or dextromethorphan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brown, Principal Investigator — NRG Oncology
Locations (220):
- United States (212):
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - SIH Cancer Institute, Carterville, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - 21st Century Oncology MHP - Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - 21st Century Oncology MHP - Farmington, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - 21st Century Oncology MHP - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Radiation Therapy-Northfield, Northfield, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - NHRMC Radiation Oncology - 16th Street, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Ogden Regional Medical Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
- Canada (8):
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Brown PD, Gondi V, Pugh S, Tome WA, Wefel JS, Armstrong TS, Bovi JA, Robinson C, Konski A, Khuntia D, Grosshans D, Benzinger TLS, Bruner D, Gilbert MR, Roberge D, Kundapur V, Devisetty K, Shah S, Usuki K, Anderson BM, Stea B, Yoon H, Li J, Laack NN, Kruser TJ, Chmura SJ, Shi W, Deshmukh S, Mehta MP, Kachnic LA; for NRG Oncology. Hippocampal Avoidance During Whole-Brain Radiotherapy Plus Memantine for Patients With Brain Metastases: Phase III Trial NRG Oncology CC001. J Clin Oncol. 2020 Apr 1;38(10):1019-1029. doi: 10.1200/JCO.19.02767. Epub 2020 Feb 14. PMID 32058845
- Available data/document: Individual Participant Data Set: NCT02360215 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Registered patients who completed required baseline neurocognitive assessments were randomized. Of 561 registered patients, 518 were randomized.
Groups:
- HA-WBRT + Memantine: Whole brain radiation therapy with hippocampal avoidance (HA-WBRT) and memantine
Period: Overall Study
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Started | 257 | 261
All Randomized Participants | 257 | 261
Started Protocol Treatment | 232 | 223
MDASI-BT Symptom Score (M.D. Anderson Symptom Inventory-Brain Module (MDASI-BT) baseline symptom severity subscale completed) | 249 | 251
MDASI-BT Intererence Score (MDSAI-BT symptom interference subscale completed at baseline) | 248 | 251
MDASI-BT Cognitive Factor Score (MDSAI-BT cognifitive factor subscale completed at baseline) | 249 | 251
MDASI-BT Neurologic Factor Score (MDSAI-BT neurologic factor subscale completed at baseline) | 249 | 251
HVLT-R Total Recall (Has standardized baseline Hopkins Verbal Learning Test - Revised (HVLT-R) Total Recall score) | 256 | 259
HVLT-R Delayed Recall (Has standardized baseline HVLT-R Delayed Recall score) | 256 | 259
HVLT-R Recognition (Has standardized baseline HVLT-R Recognition score) | 255 | 259
Trail Making Test (TMT) Part A (Has standardized baseline TMT Part A score) | 256 | 260
TMT Part B (Has standardized baseline TMT Part B score) | 250 | 257
Controlled Oral Word Association (COWA) (Has standardized baseline COWA score) | 257 | 261
Clinical Trial Battery Composite Score (Has standarized baseline Clinical Trial Battery Composite (CTB COMP) score) | 255 | 259
EQ-5D-5L Index at 2 Months (EQ-5D-5L index score completed at baseline and 2 months from treatment start) | 142 | 125
EQ-5D-5L Index at 4 Months (EQ-5D-5L index score completed at baseline and 4 months from treatment start) | 110 | 96
EQ-5D-5L Index at 6 Months (EQ-5D-5L index score completed at baseline and 6 months from treatment start) | 79 | 70
EQ-5D-5L Index at 12 Months (EQ-5D-5L index score completed at baseline and 12 months from treatment start) | 56 | 45
EQ-5D-5L VAS at 2 Months (EQ-5D-5L visual analogue scale (VAS) completed at baseline and 2 months from treatment start) | 139 | 123
EQ-5D-5L VAS at 4 Months (EQ-5D-5L visual analogue scale (VAS) completed at baseline and 4 months from treatment start) | 104 | 193
EQ-5D-5L VAS at 6 Months (EQ-5D-5L visual analogue scale (VAS) completed at baseline and 6 months from treatment start) | 76 | 69
EQ-5D-5L VAS at 12 Months (EQ-5D-5L visual analogue scale (VAS) completed at baseline and 12 months from treatment start) | 57 | 48
Completed (Subjects contributing data to results are considered to have completed the study.) | 257 | 261
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine | Total
Number analyzed (Participants) | 257 | 261 | 518
Age, Continuous [Median (Full Range); unit: years] | 61 [20 to 88] | 62 [27 to 91] | 61.5 [20 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 150 | 299
  Male | 108 | 111 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 231 | 229 | 460
  Unknown or Not Reported | 21 | 23 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 29 | 52
  White | 206 | 205 | 411
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 22 | 45
Primary tumor [Count of Participants; unit: Participants]
  Bone | 1 | 1 | 2
  Breast | 45 | 51 | 96
  Colon | 6 | 4 | 10
  Esophagus | 7 | 6 | 13
  Gastroesophageal Junction | 1 | 1 | 2
  Kidney | 8 | 5 | 13
  Lung | 151 | 156 | 307
  Ovary | 3 | 3 | 6
  Skin | 7 | 15 | 22
  Analcanal | 2 | 1 | 3
  Pancreas | 1 | 1 | 2
  Other | 25 | 17 | 42
Karnofsky Performance Status [Count of Participants; unit: Participants] — 70 = Cares for self; unable to carry on normal activity or to do active work; 80 = Normal activity with effort; some signs or symptoms of disease; 90 = Able to carry on normal activity, minor signs or symptoms of disease; 100 = Normal no complaints; no evidence of disease.
  Participants
    70 | 53 | 48 | 101
    80 | 75 | 81 | 156
    90 | 95 | 85 | 180
    100 | 34 | 47 | 81
Neurologic Function Status [Count of Participants; unit: Participants] — NS = neurologic symptoms; FA = fully active at home/work
  Participants
    No neurologic symptoms, FA without assistance | 119 | 113 | 232
    Minor neurologic symptoms, FA without assistance | 86 | 92 | 178
    Moderate NS, FA but requires assistance | 27 | 24 | 51
    Moderate NS, less than FA and requires assistance | 15 | 18 | 33
    Unknown | 9 | 13 | 22
    Not Reported | 1 | 1 | 2
Recursive Partitioning Analysis (RPA) Class [Count of Participants; unit: Participants] — The Radiation Therapy Oncology Group (RTOG) previously developed three prognostic classes for patients with brain metastases using recursive partitioning analysis (RPA) of a large database. (This study only includes the first two classes.) Class I = Karnofsky Performance Status (KPS) ≥ 70, primary controlled, age < 65, metastasis in brain only. Class II = KPS ≥ 70 and 1 of the following: primary uncontrolled; primary controlled, age ≥ 65; primary controlled, age < 65, metastases in brain & other sites.
  Participants
    Class I | 38 | 33 | 71
    Class II | 219 | 228 | 447
Prior Radiosurgery [Count of Participants; unit: Participants]
  No | 197 | 200 | 397
  Yes | 60 | 61 | 121
Prior Surgical Resection [Count of Participants; unit: Participants]
  No | 189 | 198 | 387
  Yes | 68 | 63 | 131
Metastases [Count of Participants; unit: Participants]
  Brain | 98 | 98 | 196
  Brain and Other Sites | 159 | 163 | 322
Education [Count of Participants; unit: Participants]
  No formal education | 1 | 1 | 2
  Grade school | 9 | 5 | 14
  Not high education graduate | 15 | 22 | 37
  High school graduate (including equivalency) | 86 | 85 | 171
  Some college or associate degree | 68 | 71 | 139
  Bachelor's Degree | 43 | 38 | 81
  Master's Degree | 17 | 22 | 39
  Doctoral degree or professional degree | 5 | 8 | 13
  Not reported | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to Neurocognitive Failure
Description: Neurocognitive failure is defined as the first failure, defined as a neurocognitive decline using the reliable change index (RCI) on at least one of the following assessments or parts of : Hopkins Verbal Learning Test - Revised (HVLT-R), Trail Making Test (TMT), or Controlled Oral Word Association (COWA). The HVLT-R has 3 parts that were analyzed separately for decline: Total Recall, Delayed Recall, and Delayed Recognition. The TMT has 2 parts that were analyzed separately: Part A and Part B. Neurocognitive failure rate is estimated using the cumulative incidence method. Analysis was planned to occur after 233 events were reported. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Six-month rates are provided.Analysis was planned to occur after 233 events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up was 15.6 months.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 257 | 261
percentage of participants | 68.2 [61.2 to 74.2] | 59.3 [51.9 to 66.0]
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Null hypothesis: the addition of HA-WBRT as compared to WBRT will increase time to neurocognitive failure from 53.8% in the WBRT arm to 42.8% in the HA-WBRT arm at 6 months. Treating death as a competing risk and using a Gray's test with two-sided α=0.05 to test for statistically significant difference in the distribution of neurocognitive failure times, it was calculated that 230 events over both arms would provide 90% statistical power; Test type: Superiority; p = 0.029, Gray's test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.59 to 0.96]

2. Secondary Outcome: Change From Baseline in the Hopkins Verbal Learning Test -Revised (HVLT-R) Total Recall Score (Neurocognitive Decline)
Description: The HVLT-R assesses verbal learning and memory. The test involves memorizing a list of 12 nouns for 3 consecutive trials (Total Recall), recalling the 12 targets after a 20-minute delay (Delayed Recall), and then identifying the 12 targets from a list of semantically related or unrelated items (delayed recognition). Raw scores are derived for total recall (sum of the number of targets correctly recalled), delayed recall (sum of the number of targets correctly recalled), and a delayed recognition discrimination index (sum of targets incorrectly identified subtracted from the sum of the number of targets correctly identified). The range of scores for total recall is 0 to 36, for delayed recall is 0 to 12, and -12 to 12 for recognition. A higher score indicates better functioning. Scores are standardized, adjusting for age, education, and gender as necessary, such that mean 0 and standard deviation is 1. Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with standardized score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 149 | 129
units on a scale
  2 months | -0.63 (1.25) | -0.47 (1.21)
  4 months: number analyzed (Participants) | 110 | 93
  4 months | -0.68 (1.29) | -0.36 (1.16)
  6 months: number analyzed (Participants) | 82 | 68
  6 months | -0.34 (1.33) | -0.06 (1.14)
  12 months: number analyzed (Participants) | 60 | 46
  12 months | -0.55 (1.52) | -0.34 (1.34)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Symptom Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.0586, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Symptom Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (>61 year vs. <= 61 years) is reported here; Test type: Superiority; p = 0.0048, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Symptom Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline Total Recall is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

3. Secondary Outcome: Change From Baseline in the Hopkins Verbal Learning Test -Revised (HVLT-R) Delayed Recall Score (Neurocognitive Decline)
Description: as for outcome 2
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with standardized score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 256 | 259
units on a scale
  2 months: number analyzed (Participants) | 148 | 128
  2 months | -0.75 (1.51) | -0.73 (1.53)
  4 months: number analyzed (Participants) | 109 | 93
  4 months | -0.88 (1.61) | -0.68 (1.44)
  6 months: number analyzed (Participants) | 80 | 68
  6 months | -0.54 (1.55) | -0.30 (1.31)
  12 months: number analyzed (Participants) | 60 | 46
  12 months | -0.89 (1.65) | -0.87 (1.71)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recall Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.2656, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recall Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p = 0.0067, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recall Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline Delayed Recall is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

4. Secondary Outcome: Change From Baseline in the Hopkins Verbal Learning Test -Revised (HVLT-R) Delayed Recognition (Neurocognitive Decline)
Description: The HVLT-R assesses verbal learning and memory. The test involves memorizing a list of 12 nouns for 3 consecutive trials (Total Recall), recalling the 12 targets after a 20-minute delay (Delayed Recall), and then identifying the 12 targets from a list of semantically related or unrelated items (delayed recognition). Raw scores are derived for total recall (sum of the number of targets correctly recalled), delayed recall (sum of the number of targets correctly recalled), and a delayed recognition discrimination index (sum of targets incorrectly identified subtracted from the sum of the number of targets correctly identified). The range of scores for total recall is 0 to 36, for delayed recall is 0 to 12, and -12 to 12 for recognition. A higher score indicates better functioning. Scores are standardized by expressing the deviation from the mean score of the group in units of standard deviation. Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 256 | 259
units on a scale
  2 months: number analyzed (Participants) | 148 | 126
  2 months | -0.69 (1.90) | -0.70 (1.88)
  4 months: number analyzed (Participants) | 109 | 93
  4 months | -0.11 (1.98) | -0.12 (1.41)
  6 months: number analyzed (Participants) | 80 | 68
  6 months | -0.55 (1.83) | -0.06 (1.40)
  12 months: number analyzed (Participants) | 60 | 46
  12 months | -0.48 (2.12) | -0.30 (1.65)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recognition Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.0993, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recognition Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with HVLT-R Delayed Recognition Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline Delayed Recognition is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

5. Secondary Outcome: Change From Baseline in the Trail Making Test (TMT) Part A (Neurocognitive Decline)
Description: The TMT is a neuropsychological test of visual attention and task switching that can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the first (Part A), the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order; in the second part (Part B), the subject alternates between numbers and letters (1, A, 2, B, etc.). The score is the amount of time, in seconds, that it takes the patient to complete each maze. The range for Part A is 0 to 180 (3 minutes) and for Part B is 0 to 300 (5 minutes). Lower scores indicate better functioning. Scores are standardized, adjusting for age, education, gender as needed, so that mean is 0 and standard deviation is 1. Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with standardized score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 256 | 260
units on a scale
  2 months: number analyzed (Participants) | 148 | 130
  2 months | -1.42 (6.27) | -1.31 (5.47)
  4 months: number analyzed (Participants) | 109 | 93
  4 months | -0.28 (2.42) | 0.03 (2.80)
  6 months: number analyzed (Participants) | 82 | 68
  6 months | -2.09 (13.02) | 0.17 (2.19)
  12 months: number analyzed (Participants) | 60 | 47
  12 months | -1.28 (5.10) | -0.70 (3.10)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part A (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.5988, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part A (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part A (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline TMT Part A is reported here; Test type: Superiority; p < 0.0001, McNemar; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

6. Secondary Outcome: Change From Baseline in the Trail Making Test (TMT) Part B (Neurocognitive Decline)
Description: The TMT is a neuropsychological test of visual attention and task switching that can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the first (Part A), the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order; in the second part (Part B), the subject alternates between numbers and letters (1, A, 2, B, etc.). The score is the amount of time, in seconds, that it takes the patient to complete each maze. The range for Part A is 0 to 180 (3 minutes) and for Part B is 0 to 300 (5 minutes). A lower score indicates better functioning. Scores are standardized by expressing the deviation from the mean score of the group in units of standard deviation. Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 250 | 257
units on a scale
  2 months: number analyzed (Participants) | 138 | 125
  2 months | -2.86 (16.60) | -2.27 (9.91)
  4 months: number analyzed (Participants) | 99 | 90
  4 months | -3.38 (17.88) | -0.89 (6.14)
  6 months: number analyzed (Participants) | 78 | 67
  6 months | -0.47 (7.78) | -1.06 (6.55)
  12 months: number analyzed (Participants) | 58 | 46
  12 months | -2.49 (8.18) | -1.44 (6.59)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part B (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.9226, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part B (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p < 0.0024, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with TMT Part B (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline TMT Part B is reported here; Test type: Superiority; p < 0.0001, Regression, Cox; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

7. Secondary Outcome: Change From Baseline in the Controlled Oral Word Association (COWA) Test (Neurocognitive Decline)
Description: The COWA is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter. Patients are given 1 minute to name as many words as possible beginning with the designated letter. The procedure is then repeated for the remaining two letters. Two alternate forms of the COWA are employed to minimize practice effects. The score is the sum of the correct responses with a range of 0 to infinity. A higher score indicates better functioning. Scores are standardized, adjusting for age, education, and gender as necessary, such that mean is 0 and standard deviation is 1. Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with standardized score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 257 | 261
units on a scale
  2 months: number analyzed (Participants) | 149 | 128
  2 months | -0.28 (0.96) | -0.29 (1.04)
  4 months: number analyzed (Participants) | 108 | 95
  4 months | -0.06 (0.98) | -0.08 (0.99)
  6 months: number analyzed (Participants) | 81 | 68
  6 months | -0.15 (0.87) | -0.11 (1.04)
  12 months: number analyzed (Participants) | 80 | 68
  12 months | -0.44 (1.71) | -0.21 (1.65)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with COWA (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline COWA is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with COWA (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.9749, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with COWA (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here. is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

8. Secondary Outcome: Change From Baseline in the Clinical Trial Battery Composite (CTB COMP) Score [Neurocognitive Decline]
Description: Clinical Trial Battery Composite score is the arithmetic mean of the HVLT-R (Free Recall, Delayed Recall, Delayed Recognition), TMTA, TMTB, and COWA scores, all of which are standardized, adjusting for age, education, and gender as necessary, such that mean is 0 and standard deviation is 1. A participant must have at least 5 of the 6 scores. A higher composite score indicates better neurocognitive function.Change is calculated as baseline score subtracted from post-baseline score.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with standardized score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 255 | 259
units on a scale
  2 months: number analyzed (Participants) | 148 | 127
  2 months | -1.09 (3.45) | -0.87 (2.35)
  4 months: number analyzed (Participants) | 107 | 92
  4 months | -0.81 (3.22) | -0.27 (1.66)
  6 months: number analyzed (Participants) | 80 | 68
  6 months | -0.44 (1.71) | -0.21 (1.65)
  12 months: number analyzed (Participants) | 60 | 46
  12 months | -0.98 (2.51) | -0.61 (2.00)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with the neurocognitive composite score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.2552, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with the neurocognitive composite score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with the neurocognitive composite score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline composite score is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

9. Secondary Outcome: Change in M. D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Symptom Severity Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Symptom Severity) is the average of the subscale items, given that a specified minimum numbers of items were completed.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 249 | 251
score on a scale
  2 months: number analyzed (Participants) | 146 | 126
  2 months | 0.48 (1.39) | 0.61 (1.62)
  4 months: number analyzed (Participants) | 113 | 99
  4 months | 0.29 (1.50) | 0.36 (1.46)
  6 months: number analyzed (Participants) | 81 | 71
  6 months | 0.24 (1.49) | -0.09 (1.34)
  12 months: number analyzed (Participants) | 61 | 47
  12 months | 0.53 (1.69) | 0.09 (1.47)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Symptom Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.57, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Symptom Severity score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline symptom severity is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A two-sample t-test with a 2-sided type I error of 0.05 provides >90% statistical power to detect a medium effect size of 0.5 for a comparison of the change from baseline to 6 months from the start of treatment. The comparison at six months was tested within a mixed effects model with covariates age, RPA class, prior radiosurgery, prior surgical resection, baseline score, treatment arm, and time was used; Test type: Superiority; p = 0.083, Mixed Models Analysis

10. Secondary Outcome: Change in M. D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Interference Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Interference) is the average of the subscale items, given that a specified minimum numbers of items were completed.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 248 | 251
score on a scale
  2 months: number analyzed (Participants) | 143 | 124
  2 months | 0.84 (2.45) | 1.09 (2.79)
  4 months: number analyzed (Participants) | 112 | 99
  4 months | 0.35 (2.57) | 0.51 (2.60)
  6 months: number analyzed (Participants) | 81 | 71
  6 months | 0.57 (2.61) | 0.01 (2.72)
  12 months: number analyzed (Participants) | 60 | 47
  12 months | 0.64 (2.86) | 0.14 (3.00)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Interference Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.9118, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Interference Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline interference score is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

11. Secondary Outcome: Change in M. D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Cognitive Factor Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Cognitive Factor) is the average of the subscale items, given that a specified minimum numbers of items were completed.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 249 | 251
score on a scale
  2 months: number analyzed (Participants) | 146 | 125
  2 months | 0.45 (1.81) | 0.50 (1.95)
  4 months: number analyzed (Participants) | 113 | 99
  4 months | 0.52 (1.64) | 0.32 (1.78)
  6 months: number analyzed (Participants) | 81 | 71
  6 months | 0.57 (2.61) | 0.01 (2.72)
  12 months: number analyzed (Participants) | 61 | 47
  12 months | 1.04 (2.33) | 0.50 (1.69)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Cognitive Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.1964, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Cognitive Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline cognitive factor score is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Cognitive Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Prior radiotherapy (yes vs. no) is reported here; Test type: Superiority; p = 0.0032, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

12. Secondary Outcome: Change in M. D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) Neurologic Factor Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 (best condition) to 10 (worst condition). A subscale score (Neurologic Factor) is the average of the subscale items, given that a specified minimum numbers of items were completed.
Time Frame: Baseline, 2, 4, 6, and 12 months
Population: Participants with baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 249 | 251
score on a scale
  2 months: number analyzed (Participants) | 146 | 124
  2 months | 0.17 (1.91) | 0.28 (2.31)
  4 months: number analyzed (Participants) | 113 | 99
  4 months | 0.13 (2.06) | 0.24 (1.97)
  6 months: number analyzed (Participants) | 81 | 71
  6 months | 0.23 (1.89) | 0.15 (2.11)
  12 months: number analyzed (Participants) | 61 | 47
  12 months | 0.60 (2.20) | 0.40 (2.53)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Neurologic Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Treatment Arm (WBRT+Memantine vs. HA-WBRT Memantine) is reported here; Test type: Superiority; p = 0.8877, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Neurologic Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Baseline neurologic factor is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; A mixed effects model was run with MDASI-BT Neurologic Factor Score (baseline, 2, 4, 6, and 12 months) as the outcome of interest. Age, RPA class, prior radiosurgery, prior surgical resection were the covariates considered in each model along with interaction terms treatment*time, time*time, time*time*time and remained if p<0.05. Baseline score, treatment arm, and time were forced into the model. Age (> 61 years vs. <= 61 years) is reported here; Test type: Superiority; p = 0.0078, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

13. Secondary Outcome: Change in EQ-5D-5L Index Score at 2 Months
Description: The EQ-5D-5L is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 5 problem levels (1-none to 5-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm scale ranging from 0 for the worst imaginable health state to 100 for best imaginable health state, marked at 10-point intervals. The index score is reported here.
Time Frame: Baseline and 2 months
Population: Participants with baseline and 2-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 142 | 125
score on a scale | -0.04 (0.17) | -0.05 (0.16)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.86, t-test, 2 sided — Significance level = 0.05

14. Secondary Outcome: Change in EQ-5D-5L Index Score at 4 Months
Description: as for outcome 13
Time Frame: Baseline and 4 months
Population: Participants with baseline and 4-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 110 | 96
score on a scale | -0.03 (0.17) | -0.03 (0.16)

15. Secondary Outcome: Change in EQ-5D-5L Index Score at 6 Months
Description: as for outcome 13
Time Frame: Baseline and 6 months
Population: Participants with baseline and 4-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- HA-WBRT + Memantin: Whole brain radiation therapy with hippocampal avoidance (HA-WBRT) and memantine
Arm/Group | WBRT + Memantine | HA-WBRT + Memantin
Number analyzed (Participants) | 79 | 70
score on a scale | -0.03 (0.14) | -0.03 (0.17)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantin; Test type: Superiority; p = 0.95, t-test, 2 sided — Significance level = 0.05

16. Secondary Outcome: Change in EQ-5D-5L Index Score at 12 Months
Description: as for outcome 13
Time Frame: Baseline and 12 months
Population: Participants with baseline and 12-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 56 | 45
score on a scale | -0.03 (0.17) | -0.01 (0.14)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.66, t-test, 2 sided — Significance level = 0.05

17. Secondary Outcome: Change in EQ-5D-5L VAS Score at 2 Months
Description: The EQ-5D-5L is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 5 problem levels (1-none to 5-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm scale ranging from 0 for the worst imaginable health state to 100 for best imaginable health state, marked at 10-point intervals. The VAS score is reported here.
Time Frame: Baseline and 2 months
Population: Participants with baseline and 2-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 139 | 123
score on a scale | -5.64 (24.67) | -1.41 (25.79)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.18, t-test, 2 sided — Significance level = 0.05

18. Secondary Outcome: Change in EQ-5D-5L VAS Score at 4 Months
Description: as for outcome 17
Time Frame: Baseline and 4 months
Population: Participants with baseline and 4-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 104 | 93
score on a scale | -1.35 (23.14) | -2.98 (25.71)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.64, t-test, 2 sided — Significance level = 0.05

19. Secondary Outcome: Change in EQ-5D-5L VAS Score at 6 Months
Description: as for outcome 17
Time Frame: Baseline and 6 months
Population: Participants with baseline and 6-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 76 | 69
score on a scale | 3.97 (25.33) | 3.49 (22.90)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.91, t-test, 2 sided — Significance level = 0.05

20. Secondary Outcome: Change in EQ-5D-5L VAS Score at 12 Months
Description: as for outcome 17
Time Frame: Baseline and 12 months
Population: Participants with baseline and 6-month scores
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 57 | 48
score on a scale | 2.86 (19.60) | 2.42 (23.37)
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Other; p = 0.92, t-test, 2 sided — Significance level = 0.05

21. Secondary Outcome: Intracranial Progression-Free Survival
Description: Intracranial progression-free survival time is defined as time from registration/randomization to the date of progression in the brain or death from any cause. Intracranial progression-free survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Analysis was planned to occur after 233 primary endpoint events (neurocognitive failure) were reported. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Six-month rates are provided.
Time Frame: From randomization to last follow-up. Analysis was planned to occur after 233 events were reported. Maximum follow-up was 15.6 months.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 257 | 261
percentage of participants | 43.9 [37.5 to 50.2] | 44.8 [38.5 to 51.2]
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.076, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.98 to 1.47] — Reference level = WBRT + Memantine

22. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Analysis was planned to occur after 233 primary endpoint events (neurocognitive failure) were reported. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Six-month rates are provided.
Time Frame: From randomization to last follow-up. Maximum follow-up was 15.6 months.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 257 | 261
percentage of participants | 54.9 [48.6 to 61.2] | 50.6 [44.2 to 57.0]
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.242, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.91 to 1.43] — Reference level = WBRT + Memantin

23. Secondary Outcome: Number of Patients With a Grade 3+ Adverse Event (AE) Regardless of Relationship to Treatment
Description: . Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE.
Time Frame: as for outcome 21
Population: Randomized participants who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | WBRT + Memantine | HA-WBRT + Memantine
Number analyzed (Participants) | 232 | 223
Participants | 144 | 131
Statistical Analysis 1: Comparison: WBRT + Memantine vs HA-WBRT + Memantine; Test type: Superiority; p = 0.47, Chi-squared — Two-sided p-value = 0.05

24. Other Pre Specified Outcome: Anxiety/Depression Measured Using the EQ-5D-5L
Description: An exploratory analysis, beginning with correlation coefficients, will be used to assess the association of symptom burden and anxiety/depression with neurocognitive function at each time point. The symptom burden items of interest are the "distressed (upset)", "sad", and "mood" items. From the EQ-5D-5L, the depression/anxiety item will be of interest.
Time Frame: Up to 12 months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Effect of Radiation Therapy Oncology Group (RTOG) RPA and the Diagnosis-specific Graded Prognostic Assessment (DSGPA) on Neurocognitive Function
Description: Neurocognitive function, as measured by the HVLT-R, COWA, and TMT, will be correlated with both the RTOG RPA and the DS-GPA classification systems. Baseline neurocognitive function for each test will be compared between both RPA classes using either a t-test or Wilcoxon-Mann-Whitney test, depending on the normality of the data.
Time Frame: Up to 12 months
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Effect of White Matter Injury and Hippocampal Volume on Neurocognitive Function
Description: Evaluated through MRI scans using physician-contoured and auto-contoured scores. Concordance rates will be assessed using Kappa statistics. The auto-contoured scores will be used for the remaining analyses due to the number of physicians reviewing the scans. White matter injury is measured by FLAIR volume change and is a continuous variable. Hippocampal volume is measured as a continuous variable also and both will be covariates considered in the Cox proportional hazards model to assess the impact on time to neurocognitive failure and the longitudinal modeling of neurocognitive function.
Time Frame: Up to 12 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: MDASI-BT Mood Variables
Description: The relationship between EQ-5D-5L and MDASI-BT mood variables and neurocognitive function will be assessed.
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up was 15.6 months.
Arm/Group | WBRT + Memantine | HA-WBRT + Memantin
All-Cause Mortality (participants affected / at risk) | 138/232 | 135/223
Serious Adverse Events (participants affected / at risk) | 98/232 | 106/223
Other Adverse Events (participants affected / at risk) | 214/232 | 201/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT + Memantine (N=232) | HA-WBRT + Memantin (N=223)
Anemia (Blood and lymphatic system disorders) | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac disorders - Other (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial tamponade (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2
Cushingoid (Endocrine disorders) | 0 | 1
Endocrine disorders - Other (Endocrine disorders) | 2 | 0
Blurred vision (Eye disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 4
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 6 | 9
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 12
Fever (General disorders) | 2 | 3
Flu like symptoms (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 2
General disorders and administration site conditions - Other (General disorders) | 2 | 2
Infusion related reaction (General disorders) | 1 | 0
Localized edema (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 2 | 4
Sudden death NOS (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bone infection (Infections and infestations) | 1 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Encephalitis infection (Infections and infestations) | 1 | 0
Endocarditis infective (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 2 | 2
Lung infection (Infections and infestations) | 4 | 7
Mucosal infection (Infections and infestations) | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 8 | 5
Small intestine infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 4
Wound infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
INR increased (Investigations) | 1 | 1
Investigations - Other (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 1 | 2
Weight loss (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 4
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10 | 7
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 9
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 6
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 2
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Movements involuntary (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 5 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 7 | 0
Somnolence (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 6 | 7
Delirium (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Peripheral ischemia (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 12 | 14
Vascular disorders - Other (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT + Memantine (N=232) | HA-WBRT + Memantin (N=223)
Anemia (Blood and lymphatic system disorders) | 38 | 43
Hearing impaired (Ear and labyrinth disorders) | 15 | 16
Blurred vision (Eye disorders) | 31 | 23
Abdominal pain (Gastrointestinal disorders) | 25 | 13
Constipation (Gastrointestinal disorders) | 60 | 41
Diarrhea (Gastrointestinal disorders) | 34 | 19
Dry mouth (Gastrointestinal disorders) | 21 | 18
Dysphagia (Gastrointestinal disorders) | 13 | 14
Nausea (Gastrointestinal disorders) | 105 | 89
Vomiting (Gastrointestinal disorders) | 43 | 34
Edema limbs (General disorders) | 25 | 18
Fatigue (General disorders) | 157 | 143
Gait disturbance (General disorders) | 27 | 22
Pain (General disorders) | 26 | 28
Mucosal infection (Infections and infestations) | 10 | 12
Dermatitis radiation (Injury, poisoning and procedural complications) | 18 | 11
Fall (Injury, poisoning and procedural complications) | 15 | 23
Alanine aminotransferase increased (Investigations) | 11 | 13
Alkaline phosphatase increased (Investigations) | 10 | 17
Aspartate aminotransferase increased (Investigations) | 6 | 12
Lymphocyte count decreased (Investigations) | 22 | 25
Platelet count decreased (Investigations) | 16 | 17
Weight loss (Investigations) | 44 | 31
White blood cell decreased (Investigations) | 13 | 20
Anorexia (Metabolism and nutrition disorders) | 73 | 69
Dehydration (Metabolism and nutrition disorders) | 13 | 15
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 20
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 18
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 6
Hypokalemia (Metabolism and nutrition disorders) | 21 | 18
Hyponatremia (Metabolism and nutrition disorders) | 22 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 26
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 49 | 42
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 11 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 6
Dizziness (Nervous system disorders) | 59 | 51
Dysgeusia (Nervous system disorders) | 18 | 23
Headache (Nervous system disorders) | 100 | 84
Memory impairment (Nervous system disorders) | 28 | 26
Nervous system disorders - Other (Nervous system disorders) | 13 | 7
Paresthesia (Nervous system disorders) | 16 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 17
Seizure (Nervous system disorders) | 16 | 9
Tremor (Nervous system disorders) | 12 | 18
Anxiety (Psychiatric disorders) | 23 | 17
Confusion (Psychiatric disorders) | 26 | 26
Depression (Psychiatric disorders) | 25 | 17
Insomnia (Psychiatric disorders) | 32 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 38
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 50 | 50
Alopecia (Skin and subcutaneous tissue disorders) | 70 | 54
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 6
Hypertension (Vascular disorders) | 13 | 17
Hypotension (Vascular disorders) | 10 | 12
Thromboembolic event (Vascular disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT02360215/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT02360215/ICF_001.pdf